CLINICAL TRIAL: NCT04282096
Title: Nutritional Caracterisation of Micellar Casein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ingredia S.A. (Industry)
Responsible Party: Principal Investigator, Pr Ruddy Richard, Professor, MD, PhD, Centre de Recherche en Nutrition Humaine d'Auvergne
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ID RCB 2017-A03192-51; CRNH 2017-4 (Other: Centre de Recherche en Nutrition Humaine d'Auvergne)
Record Dates: First submitted 2018-11-06; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Protein Digestion
Keywords: Micellar casein; Bioavailibility; Gastric emptying

STUDY DESIGN:
Who Masked: Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Caseine micellar (Experimental)
  Interventions: Other: native and non native casein
- Sodium Casein (Other)
  Interventions: Other: native and non native casein
- Calcium casein (Other)
  Interventions: Other: native and non native casein

INTERVENTIONS:
Other: native and non native casein — selected participant will test the 3 treatments in a random order

SUMMARY:
There are different types of casein on the market, which differ according to their chemical or physical process of obtaining. The processes will impact structural differences in the macromolecular assembly.

The majority of caseins marketed in nutrition are casein in the form of Na caseinate or Ca caseinate.

The micellar caseins obtained by membrane filtration (physical process) are more and more used in the nutrition market.

The development of casein extraction with different structures on an industrial scale opens up other perspectives for these proteins, particularly in terms of health.

The main objective of this project is to study the postprandial kinetics of the plasma concentrations of the essential amino acids of three structurally different types of caseins.

The secondary objective is to study the speed of gastric emptying and the nutritional properties of different proteins.

DETAILED DESCRIPTION:
All the participants will give freely their written informed consent before their selection in the study.

Each subject will participate in 3 kinetics of 5 hours with a different product test each time, in a randomized order. A wash-out period of at least 7 days will be respected between each kinetics. The products to be tested will be in the form of a powder (25g individual sachet, including 20.1g of protein) which will be reconstituted in 250ml of water and to which 100mg of 13C sodium acetate will be added.

For each of the kinetics, blood samples, expires gasses, will be collected at different time during the kinetics. A urinary collection throughout the day of kinetics will also be performed to allow the determination of urinary nitrogen Indirect calorimetry measurements will be performed 45 minutes every hour in the postprandial period and a measurement of 45 minutes will be made when the subject is fasting. Six measurements of indirect calorimetry will be performed for each kinetic.

Finally subjects will be asked to evaluate their satiety on a visual analog scale, 15' before taking the product, then every 15' the first hour in the postprandial period and every 30 'from the 2nd hour.

The subjects will also have a tolerance questionnaire to complete with each kinetic.

At the end of the kinetics, a standardized meal, single menu, consumption ad libitum measured in double weighing will be proposed to the volunteers to evaluate their satiety

During the 3 days preceding each kinetics, the protein intake of the subjects will be controlled. The meal of each night in the evening of kinetics will be standardized and identical for each kinetics. The volunteers will complete a food survey on the 3 days of control of their diet that precede each kinetics.

ELIGIBILITY:
Inclusion Criteria:

* - Aged 20 to 40 years
* BMI : 18.5-30 Kg/m2
* Healthy (apparently free of diseases)
* Without dietary supplement the last month
* Without allergy, lactose intolerance or aversion for milk protein
* Moderately physically active
* Affiliated to National Health Insurance
* Having provided her written informed consent

Exclusion Criteria:

* Following any kind of treatment
* Smokers (>5 cigarets/d)
* Vegetarian, vegan
* Individual unable to give informed consent or refusing to sign informed consent
* Being in exclusion on the National Volunteers Data file or refusing to be registered on the National Volunteers Data file
* Currently participating or who having got 4500€ in this year before to have participating in another clinical trial

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Changes in the plasma concentrations of the essential amino acids of 3 structurally different types of caseins during postprandial kinetics | before and during 300 minutes after product consumption
  Maximum total plasma concentration of the essential amino acids measured during different points of the 5 hours of the kinetics (one kinetic / type of casein). One point before (basal) and several points (15, 30, 45, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes) after the consumption of one of the 3 types of caseins

SECONDARY OUTCOMES:
Maximum plasma concentration for non essential amino acids | before and during 300 minutes after product consumption
  Maximum total plasma concentration of the non essential amino acids measured during different points of the 5 hours of the kinetics (one kinetic / type of casein). One point before (basal) and several points (15, 30, 45, 60, 90, 120, 150, 180, 210, 240, 270, 300 minutes) after the consumption of one of the 3 types of caseins
Tmax | before and during 300 minutes after product consumption
  Time in minutes to obtain the maximal total plasma concentration of essential amino acides
Measurement of gastric emptying by the 13C sodium acetate method | before and during 300 minutes after product consumption
  Time to obtain the maximum expired 13CO2 concentration (Tmax)
gastric emptying at 50% (T 1/2) | before and during 300 minutes after product consumption
  Obtaining time for gastric emptying at 50% (T 1/2)
Thermogenic effect of proteins at different times of kinetics | before and during 300 minutes after product consumption
  Oxidation of substrates (lipids, proteins, carbohydrates) (g/min) by indirect respiratory calorimetry corrected for nitrogen excretion.
Satietogenic effect of proteins evaluated using a visual analogue scale at different times of kinetics | from product consumption until 300 minutes after
  Measured by a visual analogue scale 100mm in length with words anchored at each end, expressing the most positive and the most negative rating, were used to assess hunger, satiety, fullness, prospective food consumption.
Tolerance of products assessed by a questionnaire | at 300 minutes after product consumption
Changes in the plasma concentrations of insulin at different times of kinetics | before and during 300 minutes after product consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche en Nutrition Humaine, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No